CLINICAL TRIAL: NCT03195296
Title: T and B Cells Infiltrating Orbital Tissues in Graves' Orbitopathy (GO) and Their Relation With GO Features
Brief Title: T and B Cells in Graves' Orbitopathy
Acronym: LYMPHGO
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Other Study IDs: LYMPHGO
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fibroadipose orbital tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graves' Orbitopathy: Patients with Graves' Orbitopathy subjected to orbital decompression
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention related to the study is foreseen

SUMMARY:
Graves orbitopathy (GO) is an inflammatory eye disease associated in 95% of patients with Graves' hyperthyroidism (GH), in ~3-4% with hypothyroid autoimmune thyroiditis, and in ~1-2% with thyroid autoimmunity in the absence of thyroid dysfunction, the former known as euthyroid GO. The pathogenesis of GO is autoimmune, with the TSH-receptor being considered the major autoantigen, thereby establishing a pathogenetic link between the thyroid and orbital tissue. Thus, TSH-receptor is expressed by orbital fibroblasts, where it forms a complex with the IGF-1 receptor. Unlike GH, which is notoriously caused by TSH-receptor stimulating autoantibodies, GO is believed to reflect cell-mediated autoimmunity, as suggested by studies showing a Th1-like pattern of cytokine release by primary cultures of orbital infiltrating lymphocytes from GO patients. On the other hand, a role of B lymphocytes has emerged in recent years based on the observation that the anti-CD20 monoclonal antibody rituximab has a beneficial effect on GO activity, as demonstrated by a recent randomized clinical trial in which rituximab was compared with intravenous glucocorticoids (GC), being the former the standard treatment of moderately-severe GO. The explanation for the findings was that B lymphocytes are involved in the pathogenesis of GO as antigen-presenting cells. However, in spite of the above mentioned promising observations, another randomized clinical trial in which rituximab was compared with placebo provided opposite results. Thus, rituximab had no effect at all on GO. Data from the two studies were confronted and major differences between the two cohorts emerged, especially concerning GO activity, leading to the conclusion that rituximab may be effective for active, but not for inactive GO. Rituximab has been employed also for autoimmune diseases other than GO, including type 1 diabetes. In the former, it was shown that the effectiveness of rituximab paralleled the presence of CD20-positive infiltrating lymphocytes in pancreas islets. We therefore postulated that something similar may occur in GO, because of which we planned the present, perspective, observational study, aimed at determining the presence and immunohistochemical features of lymphocytes infiltrating orbital tissues in patients with GO and to relate them with the clinical features of GO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Graves' orbitopathy subjected to orbital decompression

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with Graves' orbitopathy to undergo orbital decompression
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between lymphocytes infiltrating orbital tissue and GO activity | an average of 1 week
  Correlation between the number of lymphocytes infiltrating orbital tissues and the clinical activity score.
  The number of infiltrating lymphocytes is the sum of the number counted in four representative fields.
  The clinical activity score comprises 7 items (eyelid edema, conjuctival redness, eyelid redness, chemosis, caruncle edema, spontaneous eye pain, gaze-evoked eye pain), resulting in a numerical score going from 1 to 7

SECONDARY OUTCOMES:
Correlation between CD3-positive lymphocytes infiltrating orbital tissue and GO activity | an average of 1 week
  Correlation between the number of CD3-positive lymphocytes infiltrating orbital tissues and the clinical activity score.
  The number of CD3 positive infiltrating lymphocytes is the sum of the number counted in four representative fields, following immunohistochemical staining for CD3 The clinical activity score comprises 7 items (eyelid edema, conjuctival redness, eyelid redness, chemosis, caruncle edema, spontaneous eye pain, gaze-evoked eye pain), resulting in a numerical score going from 1 to 7
Correlation between CD20-positive lymphocytes infiltrating orbital tissue and GO activity | an average of 1 week
  Correlation between the number of CD20-positive lymphocytes infiltrating orbital tissues and the clinical activity score.
  The number of CD20 positive infiltrating lymphocytes is the sum of the number counted in four representative fields, following immunohistochemical staining for CD20 The clinical activity score comprises 7 items (eyelid edema, conjuctival redness, eyelid redness, chemosis, caruncle edema, spontaneous eye pain, gaze-evoked eye pain), resulting in a numerical score going from 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Michele Marinò, MD, Principal Investigator — University of Pisa

IPD SHARING:
Plan to Share IPD: No